CLINICAL TRIAL: NCT05436015
Title: Nature in Hospital - Effectiveness of Virtual Nature-based Intervention During First Stage of Labour: A Feasibility Study and Pilot RCT
Brief Title: Effectiveness of Virtual Nature-based Intervention During First Stage of Labour
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oulu (Other)
Collaborators: Oulu University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Uoulu_45/2021
Record Dates: First submitted 2022-06-13; First posted 2022-06-28 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Anxiety; Fear of Childbirth; Stress; Pain; Childbirth Experience
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial with a two-arm design will be conducted among women entering deliveryward during first stage of labour. Participants are randomized into two groups, an intervention group (N=30) and a control group (N=30). Intervention group members will receive virtual nature-based intervention; video with nature pictures and nature sounds from a 75" vertical screen monitor. Participants receive standard care during first stage of labour in both groups.
Masking Description: Statistician, who is not involved in the study has done block-randomization with variable block-sizes (2,4,6) by StatsDirect program for two groups; an intervention and control group. All study team members and participants will be blind to group allocation with the exception of one research assistant who will not be involved in providing the intervention to the participants or data analysis. Delivery ward staff (midwives) asks informed consent and after receiving it, performs the allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): In addition to usual standard care during childbirth in hospital, the intervention group will receive a virtual nature-based intervention
  Interventions: Other: Virtual nature-based intervention
- Control Group (No Intervention): The control group receives the usual standard care during childbirth in hospital

INTERVENTIONS:
Other: Virtual nature-based intervention — Virtual nature-based intervention is video with Finnish naturepictures and naturesounds shown from a 75" vertical screen monitor
  Arms: Intervention Group

SUMMARY:
Rationale: The birth environment effects on childbirth experience and feelings of security of birthing women. Fear of Childbirth (FOB) is experienced by 6-10% of women in Finland and FOB predicts postpartum depression. Real or artificial views of nature have several positive health effects including reduction of anxiety and stress. Feasible and cost-effective nature-based intervention is being studied in this pilot RCT.

Objectives: To develop a virtual nature-based intervention for the delivery ward and to assess its feasibility and effectiveness. The study assesses how the nature-based intervention carried out during the first stage of labour affects the anxiety, fear, stress, pain and childbirth experience of birthing women. The aim is to provide evidence-based information on the feasibility and effectiveness of this intervention.

Methods: Sixty women will be randomized into two groups: Nature-based intervention group and control group. All participants will have assessments during first stage of labour in nature-based intervention group before and after intervention and in control group at the same time without intervention. In both groups also 2-6 hours after childbirth, 2 days after childbirth and 2 weeks after childbirth.

DETAILED DESCRIPTION:
During the piloting and feasibility assessment phase of intervention, the nature-based intervention is tested and its feasibility and preliminary effectiveness on the anxiety, fear, stress, pain and childbirth experience is assessed. Phase II consists of a pilot RCT (Randomized Control Trial) study and a qualitative interview study. The nature-based intervention includes videos filmed in the nature of Northern Finland and takes place during 1st stage of labour before the need for medical pain relief. The pilot phase test group (N=30) will receive a nature-based intervention in addition to standard care during childbirth and the control group (N=30) receives standard care treatment. The study includes parturients (weeks of pregnancy 37+0-41+6) entering delivery ward during active labour. Before childbirth the participants in the study are measured for anxiety, stress, fear of childbirth and pain, and feeling of safety. After childbirth, the childbirth experience is assessed in the deliveryward and before discharge in postnatal ward. Before discharge, postpartum experience with anxiety, fear of childbirth and depression is also measured. During the pilot phase at two weeks, childbirth experience, anxiety and depression are assessed. Data related to childbirth and mental health diagnoses is also collected. The data is analysed using statistical methods. In the pilot phase, the participants in the intervention group (N=5-10) will be interviewed two weeks after childbirth. Thematic interview about the experiences of nature-based interventions of midwives in the delivery room (N=5-10) will also take place. Interviews are recorded and the materials are analysed by inductive content analysis.

ELIGIBILITY:
Inclusion Criteria: In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* full-term pregnancy (h 37+0 - 41+6)
* childbirth at active first-stage of labour

Exclusion Criteria: An individual who meets any of the following criteria will be excluded from participation in this study:

* severe vision or hearing loss
* communication is possible only via interpreter
* childbirth in second stage of labour
* expected complications during childbirth

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Anxiety measured with STAI-Y1, change is being assessed | 1) Pre-intervention 2) Two days after childbirth 3) Two weeks after childbirth
  The STAI meter is a two-part adult anxiety meter developed by Charles D. Spielberg and his research team (1983). It separates situation related anxiety (STATE-A = Y1) from character related tendency towards anxiety (TRAIT-A). In this study, the most used version of the STAI meter and only it's STATE-A section is utilized. Woman evaluates own current anxiety on a four-step scale with twenty questions. The respondents choose from the following options at each question: 1 = no anxiety at all, 2 = slight anxiety, 3 = some anxiety 4 = very much anxiety.

SECONDARY OUTCOMES:
1) Fear 2) Pain and 3) Feeling of Security with VAS, change is being assessed | Pre-intervention and immediately after the intervention
  VAS (Visual Analogy Scale). The VAS scale allows women to evaluate the intensity of three outcomes (three separate scales); 1) fear 2) pain and 3) feel of security on a 10cm long scale that starts at zero meaning 1) no pain 2) no fear 3) feeling of security at all and ends at 10 representing 1) the worst possible pain 2) the worst possible fear 3) the worst possible feeling of unsecurity.
Fear of Childbirth with W-DEQ version Fear of Childbirth W-DEQ version Fear of Childbirth with W-DEQ version B | Two days after childbirth
  W-DEQ version B allows women to evaluate experiences around fear of childbirth after the birth. It is currently the most widely used to measure different aspects related to the fear of childbirth. It includes 33 Likert-scale questions (0-5).
Birth Experience with NRS, change is being assessed | 1) Two - six hours after childbirth 2) two days after childbirth
  The NRS (Numeric rating scale) allows women to evaluate the birth experience from 1 to 10 immediately after birth and two days later. One means a very negative birth experience and 10 means a very positive birth experience.
Birth Experience with DSS, change is being assessed | 1) Two - six hours after childbirth 2) two days after childbirth 3) two weeks after childbirth
  The DSS (Delivery Satisfaction Scale) allows women to evaluate the birth experience with 8 questions with a 1-5 scale, 1 meaning very much and 5 not at all
Maternal Depression with EPDS, change is being assessed | 1) two days after childbirth 2) two weeks after childbirth
  EPDS (Edinburg Postnatal Depression Scale) allows women to estimate symptoms of post-natal depression. Each answer is given a score of 0 to 3 . The maximum score is 30.
Stress with physiological measures: Heart rate, change is being assessed | Pre-intervention and immediately after the intervention
  Heart rate (HR, beats per minute, BPM)
Stress with physiological measures: Heart rate variability, change is being assessed | Pre-intervention and immediately after the intervention
  Heart rate variability (HRV, milliseconds, ms)
Stress with physiological measures: Blood pressure, change is being assessed | Pre-intervention and immediately after the intervention
  Blood pressure: systolic (SBP, mmHg) and diastolic (DBP, mmHg)
Stress with physiological measures: Blood pressure variation, change is being assessed | Pre-intervention and immediately after the intervention
  Blood pressure variation (BP variation, mmHg)
Stress with physiological measures: Respiration rate, change is being assessed | Pre-intervention and immediately after the intervention
  Respiration rate (RR, breaths per minute BPM)
Stress with physiological measures: Baroreflex sensitivity, change is being assessed | Pre-intervention and immediately after the intervention
  Baroreflex sensitivity (BRS, ms/mmHg)
Stress with serum cortisol, change is being assessed | Pre-intervention and immediately after the intervention
  Serum cortisol (nmol/l)

CONTACTS AND LOCATIONS:
Overall Officials: Eila Suvanto, Study Director — Responsible investigator
Locations (1):
- Oulu University Hospital, Oulu, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aburas R, Pati D, Casanova R, Adams NG. The Influence of Nature Stimulus in Enhancing the Birth Experience. HERD. 2017 Jan;10(2):81-100. doi: 10.1177/1937586716665581. Epub 2016 Sep 30. PMID 27694185
- [Background] Berg M, Goldkuhl L, Nilsson C, Wijk H, Gyllensten H, Lindahl G, Uvnas Moberg K, Begley C. Room4Birth - the effect of an adaptable birthing room on labour and birth outcomes for nulliparous women at term with spontaneous labour start: study protocol for a randomised controlled superiority trial in Sweden. Trials. 2019 Nov 19;20(1):629. doi: 10.1186/s13063-019-3765-x. PMID 31744523
- [Background] Nielsen JH, Overgaard C. Healing architecture and Snoezelen in delivery room design: a qualitative study of women's birth experiences and patient-centeredness of care. BMC Pregnancy Childbirth. 2020 May 11;20(1):283. doi: 10.1186/s12884-020-02983-z. PMID 32393297
- [Background] Rouhe H. (2015) Fear of childbirth. Doctoral dissertation. University of Helsinki
- [Background] Ulrich, R., Simons, R., Losito, B., Fiorito, E., Miles, M., Zelson, M. (1991). Stress recovery during exposure to natural and urban environments. J. Environ. Psychol. 1991, 11, 201-230.
- [Background] Ayerle GM, Schafers R, Mattern E, Striebich S, Haastert B, Vomhof M, Icks A, Ronniger Y, Seliger G. Effects of the birthing room environment on vaginal births and client-centred outcomes for women at term planning a vaginal birth: BE-UP, a multicentre randomised controlled trial. Trials. 2018 Nov 19;19(1):641. doi: 10.1186/s13063-018-2979-7. PMID 30454075